CLINICAL TRIAL: NCT03184168
Title: A Phase 1 Open-label, Radiolabeled, Single-dose Study To Investigate The Metabolism Of [14c]Lorlatinib (Pf-06463922) In Healthy Male Volunteers
Brief Title: Single-dose Study of [14C]Lorlatinib (PF-06463922) Metabolism In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7461017; 14C ADME (Other: Alias Study Number)
Expanded Access: NCT03127618 (Approved for marketing)
Record Dates: First submitted 2017-05-17; First posted 2017-06-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers, lorlatinib, PF-06463922, ADME, NSCLC, radiolabel, metabolism
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Open-label, radiolabeled, single-dose study of an oral solution of [14C]lorlatinib (100 mg/100 µCi) in 6 healthy male volunteers. Confinement from Day -1 through Day 14 (or until 1 of 2 early release criteria is met). No returns; one follow-up phone call (at 28 to 35 days post dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): [14C]lorlatinib
  Interventions: Drug: [14C]lorlatinib

INTERVENTIONS:
Drug: [14C]lorlatinib — Extemporaneously compounded oral solution of [14C]lorlatinib (approximately 100 mg/100 µCi)
  Other Names: [14C]PF-06463922

SUMMARY:
This open-label, radiolabeled, single 100-mg dose study in 6 healthy male volunteers has been designed to further the understanding of human metabolism of lorlatinib. A prior radiolabel study using [14C]lorlatinib (study B7461004) identified an unexpected major metabolite in plasma; a benzoic acid metabolite (M8) resulting from cleavage of the amide and aromatic ether bonds of lorlatinib, accounting for 21.0% of the circulating radioactivity. However, due to the position of the 14C radiolabel on the carbonyl carbon, the metabolic fate of the larger fragment of lorlatinib resulting from this cleavage, the pyrido-pyrazole substructure, could not be determined. In this current study, the radiolabel will be on the pyrazole ring allowing for monitoring the metabolic fate of the pyrido-pyrazole part of the lorlatinib molecule cleaved during the formation of the M8 metabolite. Since M8 will not be radiolabeled, its concentrations in plasma will be determined using a validated assay.

The sample size of 6 was selected to ensure at least 4 fully evaluable subjects with completed collections of plasma, urine, and fecal samples. This is a standard sample size used for mass-balance/ADME studies which include assessment of metabolic profiling, and is not based on empirical data or hypothesis testing criteria.

Metabolic profiling of radiolabeled components will be performed on pooled plasma samples as well as on cumulative urine and feces excreted until Day 14 postdose or until one of the following early release criteria is met: 1) recovery in excreta of at least 90% of administered radioactivity, or 2) less than 1% of administered radioactivity being recovered in excreta from two consecutive days (ie, total for urine + feces should be <1% on 2 consecutive days). Plasma concentrations of both lorlatinib and its unlabeled M8 metabolite will be analyzed using validated assays. Information from this study will complement the metabolic profiling results from study B7461004, will help guide in the assessment of potential drug-drug interactions (DDIs) and the need for other DDI studies with lorlatinib.

Banked biospecimens will be collected for the purpose of conducting research. Collecting biospecimens for exploratory analyses makes it possible to better understand the investigational product's mechanism of action and to seek explanations for differences in, for example, exposure, tolerability, safety, and/or efficacy not anticipated prior to the beginning of the study.

DETAILED DESCRIPTION:
This open-label, radiolabeled, single 100-mg dose study in approximately 6 healthy male volunteers has been designed to further the understanding of human metabolism of lorlatinib. A prior radiolabel study using [14C]lorlatinib (study B7461004) identified an unexpected major metabolite in plasma; a benzoic acid metabolite (M8, PF-06895751) resulting from cleavage of the amide and aromatic ether bonds of lorlatinib, accounting for 21.0% of the circulating radioactivity or ~ 47.3% plasma M8 to lorlatinib AUC percent ratio. However, due to the position of the 14C radiolabel on the carbonyl carbon, the metabolic fate of the larger fragment of lorlatinib resulting from this cleavage, the pyrido-pyrazole substructure, could not be determined. In this current study, the radiolabel will be on the pyrazole ring allowing for monitoring the metabolic fate of the pyrido-pyrazole part of the lorlatinib molecule cleaved during the formation of the M8 metabolite. Since the M8 metabolite will not be radiolabeled, its concentrations in plasma will be determined using a validated liquid chromatography tandem mass spectrometric (LC/MS/MS) assay.

The sample size of approximately 6 was selected to ensure at least 4 fully evaluable subjects with completed collections of plasma, urine, and fecal samples. This is a standard sample size used for mass-balance/ADME studies which include assessment of metabolic profiling, and is not based on empirical data or hypothesis testing criteria.

Metabolic profiling of radiolabeled components will be performed on pooled plasma samples as well as on cumulative urine and feces excreted until Day 14 postdose or until one of the early release criteria is met. The early release criteria are: 1) recovery in excreta of at least 90% of administered radioactivity, or 2) less than 1% of administered radioactivity being recovered in excreta from two consecutive days (ie, total for urine + feces should be <1% on 2 consecutive days). Plasma concentrations of both lorlatinib and its unlabeled M8 metabolite will be analyzed using validated assays. Information from this study will complement the metabolic profiling results from study B7461004, will help guide in the assessment of potential drug-drug interactions (DDIs) and the need for other DDI studies with lorlatinib, and will aid in the understanding of the possible causes for the unexpected findings from a DDI study where a single 100 mg dose of lorlatinib was co-administered with 600 mg rifampin QD (study B7461011).

Banked biospecimens will be collected for the purpose of conducting research; specific uses are described in the Banked Biospecimens section. Comparing the deoxyribonucleic acid (DNA), ribonucleic acid (RNA), protein, and metabolite variation patterns of subjects who respond well and those who respond poorly to treatment may help to better define the most appropriate group of subjects in which to target a given treatment. Collecting biospecimens for exploratory pharmacogenomic/genomic/biomarker analyses and retaining them in the Biospecimen Banking System (BBS) make it possible to better understand the investigational product's mechanism of action and to seek explanations for differences in, for example, exposure, tolerability, safety, and/or efficacy not anticipated prior to the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (no clinically relevant abnormalities) males, 18 to 55 years at the time of screening.
2. BMI of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, CV, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding seasonal allergies).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug test.
4. History of regular alcohol consumption exceeding 14 drinks/week within 6 months before screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the dose of investigational product (whichever is longer).
6. Screening BP ≥ 140 mm Hg (systolic) or 90 mm Hg (diastolic) following at least 5 minutes of rest. If systolic or diastolic BP is higher at screening, repeat 2 times and use average of 3 BP values.
7. Screening supine 12 lead ECG QTc interval >450 msec or QRS interval >120 msec, or PR interval > 180 msec. If QTc or QRS exceed, ECG should be repeated 2 more times and the average of the 3 QTc or QRS should be used.
8. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening (and confirmed with single repeat): AST or ALT level > 1.0 × ULN; Total bilirubin level > 1.5 × ULN. If history of Gilbert's syndrome, subject would be eligible provided the direct bilirubin level is ≤ ULN.
9. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to study drug dose. Acetaminophen may be used at dosed up to 1 g/day. Limited use of nonRx medications may be permitted following approval by the sponsor. Herbal supplements and hormone replacement therapy must have been discontinued at least 28 days prior to study drug dose.
10. Blood donation (excluding plasma) of ~ 1 pint (500 mL) or more within 60 days prior to dosing.
11. History of HIV, hepatitis B, or hepatitis C; positive testing for HIV, HepBsAg, HepBcAb, or HCVAb.
12. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section.
13. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
14. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.
15. History of irregular bowel movements eg, regular episodes of diarrhea or constipation, irritable bowel syndrome or lactose intolerance.
16. Enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry (ie, occupational exposure of 5 rem per year).
17. Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.
18. Subjects who have used tobacco within 90 days prior to dosing.
19. Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Metabolic profiling for lorlatinib will be determined in plasma, urine and fecal samples. | Assessments will be made up to 14 days post dose
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces.

SECONDARY OUTCOMES:
Maximum exposure in plasma will be determined for lorlatinib, M8 metabolite and total radioactivity | Assessments will be made up to 14 days postdose
  Cmax (maximum observed plasma concentration) will be reported directly from each analyte's data
Time of maximum exposure in plasma will be determined for lorlatinib, M8 metabolite and total radioactivity | Assessments will be made up to 14 days post dose
  Tmax (Time of Cmax) will be reported directly from each analyte's data as time of first Cmax occurrence
Exposure up to the last quantifiable concentration will be determined for lorlatinib, M8 metabolite and total radioactivity | Assessments will be made up to 14 days post dose
  AUClast (Area under the plasma concentration time profile from time 0 to the time of the last quantifiable concentration) will be determined, using Linear/Log trapezoidal method, from plasma concentration data for each analyte
The overall exposure in plasma will be determined for lorlatinib, M8 metabolite and total radioactivity | Assessments will be made up to 14 days post dose
  AUCinf (Area under the plasma concentration time profile from time 0 extrapolated to infinite time) will be determined, using Linear/Log trapezoidal method, from plasma concentration data for each analyte
The terminal elimination half life in plasma will be estimated from plasma profiles over time for lorlatinib, M8 metabolite and total radioactivity | Assessments will be made up to 14 days post dose
  t1/2 (apparent terminal elimination half life) will be estimated for each analyte from the terminal portion of its plasma concentration versus time plot

OTHER OUTCOMES:
Relative routes of excretion of total radioactivity | Assessments will be made up to 14 days post dose
  Recovery (as % administered dose) of total radioactivity in urine and feces.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7461017&StudyName=A+Phase+1+Open-label%2C+Radiolabeled%2C+Single-dose+Study+To+Investigate+The+Metabolism+Of+%5B14c%5Dlorlatinib+%28pf-06463922%29+In+Healthy+Male+Volunteers